CLINICAL TRIAL: NCT01118338
Title: A Study to Evaluate the Product Performance of Two Different Designs of Bausch & Lomb PureVision® Contact Lenses
Brief Title: Evaluation of Two Different Designs of Bausch & Lomb Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 648
Record Dates: First submitted 2010-04-30; First posted 2010-05-06 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Myopia
Keywords: contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Redesigned Purevision Contact Lens (Experimental): Redesigned Bausch & Lomb PureVision contact lens
  Interventions: Device: Redesigned Purevision Contact Lens
- PureVision Contact Lens (Active Comparator): Bausch & Lomb PureVision contact lens
  Interventions: Device: PureVision Contact Lens

INTERVENTIONS:
Device: Redesigned Purevision Contact Lens — Lenses will be dispensed at screening visit, subjects will wear lenses on a daily wear basis for one month.
  Arms: Redesigned Purevision Contact Lens
Device: PureVision Contact Lens — Lenses will be dispensed at screening visit, subjects will wear lenses on a daily wear basis for one month.
  Arms: PureVision Contact Lens

SUMMARY:
The objective of this one month study is to evaluate the product performance of a redesigned PureVision Contact Lens compared to the PureVision Contact Lens when worn on a daily wear basis by wearers of contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be adapted wearers of one of the listed contact lenses
* Subjects must be myopic
* Subjects must use a lens care system on a regular basis.

Exclusion Criteria:

* Subjects who have worn gas permeable (GP) contact lenses within the last 30 days of polymethylmethacrylate (PMMA) lenses within the last 3 months.
* Subjects with any systemic disease affecting ocular health.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or are using any ocular medication.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects who have had any corneal surgery (eg, refractive surgery).
* Subjects who have participated in any drug or device clinical investigation within two weeks prior to entry into this study and/or during the period of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cairns, MCOptom, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 188 participants enrolled into each group, for a total of 376 participants enrolled. There were 185 participants in the redesigned group and 183 participants in the control group who were eligible and dispensed lenses.
Period: Overall Study
Arm/Group | Redesigned Purevision Contact Lens | PureVision Contact Lens
Started | 185 | 183
Completed | 182 | 174
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Redesigned Purevision Contact Lens | PureVision Contact Lens | Total
Number analyzed (Participants) | 185 | 183 | 368
Age, Continuous [Mean (Full Range); unit: years] | 32.0 [18 to 63] | 30.6 [18 to 52] | 31.3 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 130 | 266
  Male | 49 | 53 | 102

OUTCOME MEASURES:

1. Primary Outcome: Symptoms and Complaints
Description: Symptoms/complaints were assessed on a scale from 0 to 100, with 0 denoting unfavorable symptoms/complaints and 100 denoting the most favorable rating. The generic scale was comprised of 14 separate questions, where each assessed the denoted symptom/complaint with a score between 0 and 100. The total score was not calculated.
Time Frame: 1 month
Population: There were 185 participants (370 eyes) in the redesigned group and 183 participants (366 eyes) in the control group who were eligible and dispensed lenses. There were 368 dispensed eyes in the redesigned group and 360 dispensed eyes in the control group evaluable for the analysis population for the assessment of symptoms and complaints.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Redesigned Purevision Contact Lens | PureVision Contact Lens
Number analyzed (Participants) | 184 | 180
Number analyzed (eyes) | 368 | 360
score on a scale
  Lens handling upon insertion | 83.2 (17.7) | 83.6 (17.7)
  Comfort upon insertion | 78.1 (21.7) | 74.6 (21.7)
  Burning/stinging upon insertion | 84.6 (19.0) | 83.2 (19.0)
  Comfort throughout the day | 75.1 (22.2) | 73.0 (22.2)
  End of day comfort | 67.6 (24.8) | 65.1 (24.9)
  Lens awareness | 76.4 (22.6) | 72.1 (22.6)
  Lens cleanliness | 84.5 (16.5) | 81.5 (16.5)
  Irritation | 76.6 (22.4) | 73.4 (22.4)
  Itching | 85.7 (18.5) | 85.2 (18.5)
  Dryness | 75.1 (23.8) | 73.5 (23.9)
  Redness | 88.5 (17.6) | 86.6 (17.6)
  Vision | 82.9 (19.7) | 82.0 (19.7)
  Lens handling upon removal | 88.3 (15.5) | 86.6 (15.5)
  Overall impression | 72.8 (24.7) | 67.7 (24.7)

2. Secondary Outcome: Visual Acuity
Description: Visual acuity was assessed by distance high contrast logarithm of the minimum angle of resolution (logMAR).
Time Frame: 1 month
Population: There were 185 participants (370 eyes) in the redesigned group and 183 participants (366 eyes) in the control group who were eligible and dispensed lenses.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Redesigned Purevision Contact Lens | PureVision Contact Lens
Number analyzed (Participants) | 185 | 183
Number analyzed (eyes) | 370 | 366
logMAR | -0.028 (0.068) | -0.021 (0.068)

3. Secondary Outcome: Percentage of Eyes With > Grade 2 Slit Lamp Findings
Description: Graded slit lamp findings for each eye, including epithelial edema, epithelial microcysts, corneal staining, limbal and bulbar injections, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates were graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). The outcome measure is any finding > grade 2, across abnormalities.
Time Frame: 1 month
Population: There were 188 participants (376 eyes) enrolled into each group, for a total of 376 participants enrolled (752 eyes). There were 372 eyes in the redesigned group and 374 eyes in the control group assessed for slit lamp findings during the study.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Redesigned Purevision Contact Lens | PureVision Contact Lens
Number analyzed (Participants) | 186 | 187
Number analyzed (eyes) | 372 | 374
eyes | 5 | 5

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable. There were 376 eyes dispensed the test lens and 376 eyes dispensed the control lens, assessed for adverse events.
Arm/Group | Redesigned Purevision Contact Lens | PureVision Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/183
Other Adverse Events (participants affected / at risk) | 0/185 | 0/183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.